CLINICAL TRIAL: NCT07229989
Title: Effectiveness of a Pregnancy Care App on Maternal Knowledge and Anxiety in Pregnant Women: Quasi-Experimental Study
Brief Title: Effectiveness of a Pregnancy Care App on Maternal Knowledge and Anxiety in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lincoln University College Malaysia (Other)
Responsible Party: Principal Investigator, Nurul Jannah, M.Tr.Keb, Principle Investigator, Lincoln University College Malaysia
Organization: Lincoln University College (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUC_02_Jannah; LUC_02_Jannah (Other: Lincoln University College Malaysia)
Record Dates: First submitted 2025-09-29; First posted 2025-11-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy
Keywords: antenatal care; Prenatal education; Digital health intervention
MeSH Terms: interventions — Prenatal Care; Amyloid; Telemedicine; Pregnancy

STUDY DESIGN:
Intervention Model Description: This study uses a quasi-experimental design with a pre-test and post-test approach. Participants are assigned to one of two groups: an intervention group using the Pregnancy Care app for 21 day, and a control group receiving standard education. The study aims to evaluate the app's effectiveness in improving maternal knowledge and reducing anxiety before childbirth.
Masking Description: This study does not involve masking or blinding. All participants and investigators are aware of the group assignments and the intervention being used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Arm Type: Experimental Arm Name: Intervention Group Description: Participants in this group will use the pcycare digital for 21 day The app includes educational content and holistic therapy.
  Interventions: Behavioral: PcyCare (Pregnancy Care) App
- control group (No Intervention): Arm Type: Active Comparator Arm Name: Control Group Description: Participants in this group will receive standard maternal education without using the mobile application.

INTERVENTIONS:
Behavioral: PcyCare (Pregnancy Care) App — The Pregnancy Care App is a mobile-based self-learning platform designed to improve maternal knowledge and reduce anxiety before childbirth. It includes educational modules on pregnancy and labor preparation, as well as holistic therapy features such as antenatal yoga, acupressure, guided relaxation, meditation, self-hypnosis, mindfulness, deep breathing, journaling, and hope-based affirmations. Participants in the intervention group will use the app for two week.
  Other Names: Mobile Health for Maternal Education; Digital Holistic Therapy for Pregnancy
  Arms: Intervention Group

SUMMARY:
1. Objective:

   To evaluate the effectiveness of the Pregnancy Care mobile application in improving maternal knowledge and reducing anxiety in preparation for childbirth, through an educational and holistic therapy-based approach.
2. Key Questions:

   1. Can the Pregnancy Care app improve pregnant women's knowledge about pregnancy and childbirth preparation?
   2. Is the app effective in reducing anxiety levels among pregnant women before delivery?
   3. What are the changes in knowledge and anxiety levels before and after the intervention in the group using the app compared to the control group?
3. Procedure:

This study uses a quasi-experimental design with a pre-test and post-test approach involving two groups:

1. Intervention group: Participants will use the Pregnancy Care app for one week. The app includes educational content on physical and emotional changes during pregnancy, nutritional and activity needs, and childbirth preparation. It also features holistic therapy components such as antenatal yoga, acupressure, guided relaxation, meditation, self-hypnosis, mindfulness, deep breathing, journaling, and hope-based affirmations.
2. Control group: Participants will receive standard education without using the app.

Measurements will be taken before and after the intervention using validated questionnaires to assess knowledge and anxiety levels. The data will be analyzed to determine the effectiveness of the app in enhancing maternal readiness for childbirth

DETAILED DESCRIPTION:
Background:

Anxiety before childbirth is a common issue among pregnant women and can negatively affect the delivery process and maternal-infant health. Adequate knowledge and psychological support are essential to help mothers feel more prepared and confident.

Study Purpose:

To develop and evaluate the Pregnancy Care mobile application as a digital intervention aimed at improving maternal knowledge and reducing anxiety through educational content and holistic therapy.

App Content: The Pregnancy Care app integrates:

Educational modules covering:

Physical and emotional changes during pregnancy Nutritional and activity needs Stages of labor and delivery Pain management and breathing techniques Postpartum care and breastfeeding

Holistic therapy features:

Body: Antenatal yoga, acupressure, massage points Mind: Guided relaxation, meditation, self-hypnosis, mindfulness, deep breathing Soul: hope affirmations, spiritual and motivational content

Study Design:

A quasi-experimental design with two groups:

Intervention group: Uses the pcycare for 21 day Control group: Receives standard education without the pcycare

Measurement and Analysis:

Pre-test and post-test assessments are conducted using validated questionnaires to measure maternal knowledge and anxiety levels. Data are analyzed to determine the effectiveness of the app in improving childbirth preparedness.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged 20-40 years
2. Gestational age between 28 and 35 weeks
3. Able to read and understand the language used in the PcyCare platform
4. Owns a smartphone, tablet, or computer with internet access
5. Provides informed consent to participate

Exclusion Criteria:

1. High-risk pregnancy requiring intensive medical care
2. Severe psychiatric or cognitive disorders that would prevent platform use
3. Participation in another conflicting educational or intervention study

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2025-09-18 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Change in maternal knowledge about pregnancy care | 21 days interventions
  Maternal knowledge about pregnancy care will be evaluated as a primary outcome in this study. The assessment will utilize the Pregnancy Knowledge Questionnaire (TPKQ):, a structured instrument consisting of 10 multiple-choice questions that cover essential topics such as nutrition during pregnancy, recognition of danger signs, antenatal care practices, and birth preparedness. Each correct answer is scored as 1, while incorrect answers receive a score of 0, resulting in a total score range of 0 to 10.
  The questionnaire has been tested for validity, with a Pearson correlation coefficient (r) > 0.361, indicating all items are valid. Reliability testing using Cronbach's Alpha yielded 0.81, confirming that the instrument is highly reliable.

SECONDARY OUTCOMES:
Change in maternal anxiety levels during pregnancy | Baseline and 21 days intervention
  Maternal anxiety during pregnancy will be assessed using the Late Pregnancy Anxiety Scale (LPAS-ID) questionnaire, consisting of 8 items measured on a 4-point Likert scale (1 = Never, 2 = Rarely, 3 = Often, 4 = Very Often), resulting in a total score range of 8 to 32. The PRAS questionnaire demonstrated good validity (r > 0.361) and high reliability (Cronbach's Alpha = 0.85).
Change in birth preparedness among pregnant women | 21 days intervention
  Birth preparedness will be assessed using the Childbirth Readiness Questionnaire (CRQ), a 8-item questionnaire rated on a 4-point Likert scale (1 = Never, 2 = Rarely, 3 = Often, 4 = Very Often) with total scores ranging from 8 to 32. This instrument assesses the physical, mental, and informational readiness of pregnant women for childbirth.
  The CRQ questionnaire has strong validity (r > 0.361) and excellent reliability (Cronbach's Alpha = 0.82).

CONTACTS AND LOCATIONS:
Overall Officials: Nurul Jannah, M.Tr.Keb, Principal Investigator — Lincoln University College Malaysia
Locations (1):
- Disctrict, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected during this study will not be shared with other researchers outside the study team. This decision is based on considerations of participant confidentiality, ethical approval limitations, and the scope of the current research. All data will be used solely for the purposes of this study and will remain under the control of the principal investigator and affiliated institution.